CLINICAL TRIAL: NCT03287596
Title: Cartography and Quantitative Characterization of Achilles Tendon Fibrocartilage by TE = 0ms Imaging at3T MRI
Brief Title: Cartography and Quantitative Characterization of Achilles Tendon Fibrocartilage by TE = 0ms Imaging at 3T MRI
Acronym: SILENZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2015/16
Record Dates: First submitted 2017-09-12; First posted 2017-09-19 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Spondyloarthropathy; Tendinopathy
Keywords: Spondylarthropathy; Tendinopathy; MRI; Healthy Volunteer
MeSH Terms: conditions — Spondylarthropathies; Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HEALTHY VOLUNTEERS (Experimental): * 3D sequence ZTE2 DP without gadolinium
  * 3D Sequence UTE without gadolinium
  Interventions: Device: MRI ZTE2 sequence
- SPA + NON-SYMPTOMATICS (Experimental): * 3D sequence ZTE2 DP without gadolinium
  * 3D Sequence UTE without gadolinium
  * 3D Sequence ZTE2 DP with gadolinium
  * 3D sequence UTE with gadolinium
  Interventions: Device: MRI ZTE2 sequence
- SPA + SYMPTOMATICS (Experimental): * 3D sequence ZTE2 DP without gadolinium
  * 3D Sequence UTE without gadolinium
  * 3D Sequence ZTE2 DP with gadolinium
  * 3D sequence UTE with gadolinium
  Interventions: Device: MRI ZTE2 sequence
- MECHANIC TENDINOPATHY (Experimental): * 3D sequence ZTE2 DP without gadolinium
  * 3D Sequence UTE without gadolinium
  * 3D Sequence ZTE2 DP with gadolinium
  * 3D sequence UTE with gadolinium
  Interventions: Device: MRI ZTE2 sequence

INTERVENTIONS:
Device: MRI ZTE2 sequence — feasibility of ZTE 2 sequence to quantitatively assess normal and pathological spondyloarthropathy

SUMMARY:
The purpose of this study is to accurately map calcaneal fibrocartilage using TE = 0 ms imaging, and then apply measurements of our control population to SpA patients with peripheral enthesis study using the calcaneal tendon as a clinical model

DETAILED DESCRIPTION:
The human body contains a lot of tissue components with short T2 (transversal relaxation time) that are not or only poorly detected on conventional T2-weighted MR sequences. These components are mostly located in musculoskeletal organs such as tendons, ligaments, menisci, periosteum or cortical bone.

Considering that conventional sequences do not detect tissue components with T2 shorter than 10ms, imaging of body tendon or enthesis is therefore very limited. This represents a limitation of MR imaging in early diagnosis of a certain number of pathologies, such as mechanical or mostly inflammatory tendinopathy or enthesopathy.

This study, would provide the feasibility of ZTE 2 sequence to quantitatively assess normal and pathological spondyloarthropathy Achilles tendon enthesis at 3 T, and would demonstrate that this sequence allows the detection of SpA enthesopathy prior to conventional sequences and enables disease monitoring.

For those purposes, during inclusion visit sequences ZTE 2 and UTE (with and without gadolinium injection) will be add to routine macrocyclic gadolinium injected MRI of 3 groups of patients (symptomatic and non sympatomatic spondyloarthropathy and mechanical tendinopathy). Healthy volunteer group will undergo an MRI exam without gadolinium injection comprised of following sequences T2 FS, T1, DP FS, ZTE 2 and UTE.

No follow up visit are schedule in this study

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years,
* Covered under social security
* Informed signed consent

Additional criteria for each group:

GROUP 1: HEALTHY VOLUNTEERS

* Absence of diagnosis of spondyloarthropathies
* No previous history of plantar support and pain, calcaneal tendinopathy, infiltration or surgery

GROUP 2: SPA + NON-SYMPTOMATICS AT THE CALCANEEN FIBROCARTILAGE LEVEL

* ASAS criteria axial or appendicular
* No previous history of plantar support and pain, infiltration or surgery
* Prescription Achile's tendon MRI with injection of contrast agent (macrocyclic gadolinium) in usual care.

GROUP 3: SPA + SYMPTOMATICS AT THE CALCANEEN FIBROCARTILAGE LEVEL

* ASAS criteria axial or appendicular
* Clinical suspicion of rheumatic enthesopathy
* Absence of a history of calcaneal infiltration or surgery
* Prescription Achile's tendon MRI with injection of contrast agent (macrocyclic gadolinium) in usual care.

GROUP 4: MECHANIC TENDINOPATHY

* Clinical diagnosis of calcaneal mechanical tendinopathy
* Absence of diagnosis of spondyloarthropathies
* No any previous history of plantar support disorder, calcaneal infiltration or surgery
* Prescription Achile's tendon MRI with injection of contrast agent (macrocyclic gadolinium) in usual care.

Exclusion Criteria:

* Age less than 18 yrs old
* Pregnant or lactating woman
* History or presence coronary pathology
* Septic arthritis
* Immunodeficiency.
* Contra-indication for MRI exam
* Legal protection

Additional criteria for GROUPS 2, 3 and 4:

* History or presence of renal insufficiency
* Allergy to macrocyclic gadolinium

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
Maximum ZTE signal value in healthy volunteers | baseline

SECONDARY OUTCOMES:
Maximum difference of the ZTE signal value between healthy volunteers and non-symptomatic SpA + patients in the calcaneal fibrocartilage | baseline
Maximum difference of the ZTE signal value between healthy volunteers and symptomatic SpA + patients in the calcaneal fibrocartilage | baseline
Maximum difference in the ZTE signal value between healthy volunteers and patients with mechanical tendinopathy | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hauger, MD, Ph.D, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France